CLINICAL TRIAL: NCT01873807
Title: An Open-label,Multi-center,Prospective Study of Idarubicin and Etoposide Intensified Conditioning Regimen Allogeneic Hematopoietic Stem Cell Transplantation for Adult Acute Lymphoblastic Leukemia
Brief Title: HD-Idarubicin/Etoposide Intensified Conditioning Regimen Allo-HSCT for Adult ALL
Acronym: HITA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIE-ALL-2013
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Idarubicin; Etoposide; HSCT; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Idarubicin; Whole-Body Irradiation; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDA-Etoposide Intensified Conditioning (Experimental)
  Interventions: Drug: IDA; Radiation: TBI; Drug: CTX; Drug: VP-16
- Non-IDA Conditioning (Active Comparator)
  Interventions: Radiation: TBI; Drug: CTX; Drug: VP-16

INTERVENTIONS:
Drug: IDA — Idarubicin: 15mg/m2/d: -8->-6d
  Other Names: Idarubicin
  Arms: IDA-Etoposide Intensified Conditioning
Radiation: TBI — TBI: 4.5 Gy/d, -5d, -4d
  Other Names: Total Body Irradiation
Drug: CTX — CY:60mg/kg/d, -3d, -2d
  Other Names: Cyclophosphamide
Drug: VP-16 — VP-16: 15mg/kg, -2d, -1d
  Other Names: Etoposide

SUMMARY:
Intensified conditioning regimen allo-HSCT is based on a hypothesis of that intensifying condition with less-used drugs could overcome resistance,reduce tumor burden, and most importantly, spare enough time for slow-growing GVL effect following immune reconstitution to finally get rid of MRD and control the disease. Our previous trial of HDE-ALL-2011 (NCT01457040) have confirmed the role of intensified conditioning allo-HSCT in adult ALL, resulting in significantly improved OS and EFS in comparison with previous standard TBI/CY2 conditioning regimen(data not yet published). But at the same time, FA-TBI/CY2-VP16 conditioning regimen was associated with high transplantation-related mortality (TRM), which might be attributed to excessive suppression on both bone marrow and immune. TT-ALL-HIE-2013, substituting FA with idarubicin, is aimed at maintaining anti-tumor effect with less cross-resistance and immune suppression and reducing TRM.

DETAILED DESCRIPTION:
It's well-known that the long-term outcome of adult acute lymphoblastic leukemia (ALL) lags far behind that of pediatric ALL,associated with different molecular cytogenetics make-up and treatment strategies. In search of an optimal regimen for pediatric ALL, comprehensive series of clinical trials of intensive chemotherapies have been conducted and lead to 80%-90% long-term survival. At the same time, pediatric-inspired chemotherapy protocol aslo yielded a charming result of 50-60% 3-year EFS in adolescent and young adult. In comparison with the leading role of intensive chemotherapy in pediatric ALL, allogeneic hematopoietic stem cell transplantation (allo-HSCT) plays an important role in treatment strategy of adult ALL. According to the state-of-art understanding of ALL, total therapy of ALL should consist of molecular-cytogenetics classification at diagnosis, minimal residual disease (MRD) monitoring and redefining risk classification during treatment, pediatric-inspired chemotherapy with high-dose Methotrexate/L-asparaginase during consolidation therapy,furthermore,risk/MRD-adapted allo-HSCT for high-risk and refractory/relapsed ALL.In pre-pediatric-inspired protocol era, allo-HSCT still represents the major role for improving the outcome of adult ALL, especially for high-risk and refractory/relapsed ALL. It's established that graft-versus-leukemia (GVL) effect was weak in ALL and patient shows poor response for donor-lymphocyte infusion (DLI). Intensified conditioning regimen allo-HSCT is based on a hypothesis of that intensifying condition with less-used drugs could overcome resistance,reduce tumor burden, and most importantly, spare enough time for slow-growing GVL effect following immune reconstitution to finally get rid of MRD and control the disease. Our previous trial of HDE-ALL-2011 (NCT01457040) have confirmed the role of intensified conditioning allo-HSCT in adult ALL, resulting in significantly improved OS and EFS in comparison with previous standard TBI/CY2 conditioning regimen(data not yet published). But at the same time, FA-TBI/CY2-VP16 conditioning regimen was associated with high transplantation-related mortality (TRM), which might be attributed to excessive suppression on both bone marrow and immune. TT-ALL-HIE-2013, substituting FA with idarubicin, is aimed at maintaining anti-tumor effect with less cross-resistance and immune suppression and reducing TRM.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 16 years to 65 years;
2. Diagnosis of acute lymphoblastic leukemia;
3. Patient receives allo-HSCT;
4. The informed consent form has been signed;

Exclusion Criteria:

1. Patient with severe cardiac dysfunction with less than 50% EF;
2. Patient with severe lung dysfunction;
3. Patient with more than 3 times ULN of serum ALT or AST levels, or with more than 2 times ULN of serum TBIL level, or less than 40% of normal prothrombin time activity (PTA); or with more than 2 times the ULN of serum Cr;
4. Patient with severe active infection;
5. Patient with allergy history about suspected drug in conditioning regimen;
6. Patient with other conditions considered unsuitable for the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival | 3 year

SECONDARY OUTCOMES:
Transplantation-Related Mortality | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Department of Hematologym, Nanfang Hospital, Southern Medical University, China
Locations (13):
- China (13):
  - Department of Hematology, Union Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangdong No.2 Provincial People's Hospital, Guangzhou, Guangdong
  - Department of Hematology, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Department of Hematology, 1st Guangzhou People Hospital, Guangzhou, Guangdong
  - Oncology-Hematology Center, 1st Affiliated Hospital, Guangzhou Medical Collgege, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Zhongshan People Hospital,Guangdong, Zhongshan, Guangdong
  - Department of Hematology, 1st Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Department of Hematology, Union Hospital, Huazhong Science and Technology, Wuhan, Hubei
  - Department of Hematology, Tongji Hospital, Huazhong Science and Technology, Wuhan, Hubei

REFERENCES:
- See also: Website of Nanfang Hospital, Southern Medical University, Guangzhou, 510515, China. — http://www.nfyy.com